CLINICAL TRIAL: NCT07265687
Title: Pelvic Functional Magnetic Stimulation on Pain in Endometriosis Patients - a Prospective Non Randomised, Non-blinded Single Centre Observational Trial
Brief Title: Impact of Magnetic Stimulation on Pain in Endometriosis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tesla-Endom; 2025-D0011 (Other: Cantonal Ethics Committee Zurich)
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tesla-Chair (Experimental)
  Interventions: Device: Magnetic stimulation

INTERVENTIONS:
Device: Magnetic stimulation — Magnetic stimulation using the Tesla-Chair

SUMMARY:
Many women with endometriosis still experience pain despite surgical and medical treatment. Over-the-counter painkillers are usually helpful in alleviating this pain. But for some patients, these medications eventually stop working. Pain then dominates their daily life. In this study, we are investigating the effects of magnetic stimulation using the "Tesla chair" and whether it can alleviate their pain

DETAILED DESCRIPTION:
Patients who are diagnosed with CPP and hypertonic pelvic floor as assessed in gynaecological exam will be asked to participate. Before start of the Tesla chair treatment VAS Score by PPAF will be assessed. After 6 treatments (after 3 weeks an intermediate doctor's consultation will rule out aggravation of CPP by treatment and if possible the next cycle of 6 treatments will be scheduled. After completion of 12 treatments the VAS Score will be reassessed and treatments' success evaluated in a doctor's consultation. We plan to re-evaluate sustaining success after 3 months after treatments completion

ELIGIBILITY:
Inclusion Criteria:

* Patient has been informed about study
* Age ≥ 18 years
* Premenopausal
* histologically or laparoscopically or MRI confirmed endometriosis
* CPP (cyclical pelvic pain VAS ≥ 5)
* Pelvic floor hypertonicity
* Written informed consent
* sufficient German speaking
* Current endocrine therapy for >= 3 months

Exclusion Criteria:

* Contraindications according manufactureres manual Tesla Chair
* Pregnancy or desire to become pregnant within the next 8 weeks
* Pelvic organ prolapses
* Genital infections
* Menstruation
* active malignancy, Malignant tumors
* Severe neurological diseases
* Cardiac arrhythmia
* Active internal medical devices e.g. cardiac pacemakers, medication, pumps etc.
* Ferromagnetic implants at or near the site of stimulation
* Recent surgery at the site of stimulation
* Thrombosis or thrombophlebitis
* Epilepsy or suspected epilepsy
* Acute stages of kidney stones
* Gastrointestinal and internal disease at the site of stimulation
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* Previous enrolment into the current investigation
* Enrolment of the Sponsor or PI, their family members, employees and other dependent persons
* No endocrine therapy or use of endocrine therapy for < 3 months
* active inflammatory diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Decrease of PPAF-Score before and after treatment. | From enrollment to the end of tratment at end of week 7
  Relief of pain measured by changes in PPAF (Pelvic pain assessment form) score before and after the treatment. 0= no pain, 10 = unbearable pain

SECONDARY OUTCOMES:
Decrease of PPAF-Score before and after treatment. | From enrollment to 3 months after completion of treatment
  Relief of pain measured by changes in PPAF (Pelvic pain assessment form) score before and after the treatment. 0= no pain, 10 = unbearable pain

OTHER OUTCOMES:
Subjective experience of patients, decrease in analgetic use | From enrollment to 3 months after completion of treatment
  Subjective experience of patients, decrease in analgetic use, subjective success

IPD SHARING:
Plan to Share IPD: No